CLINICAL TRIAL: NCT01547013
Title: Phase II The Use of Near Infrared Spectroscopy in the Diagnosis of Acute Compartment Syndrome in Trauma Patients
Brief Title: The Use of Near Infrared Spectroscopy in the Diagnosis of Acute Compartment Syndrome in Trauma Patients
Acronym: NIRS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: S-11-20; A-15808.2 (Other: HRPO); I100543 (Other: FDA)
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Anterior Tibial Compartment Syndrome
MeSH Terms: conditions — Anterior Compartment Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- COHORT 1: Critical Controls: Twenty five (25) critically injured subjects with NO "severe" traumatic lower extremity traumatic injuries to provide control data for critically injured physiological status, a state which may induce systemic, vs. regional hypoperfusion. ("Critical" CONTROLS)
- COHORT 2: Ninety five (95) total (35 Cohort 2A; 35 Cohort 2B; 25 Cohort 2C) subjects with "severe leg injuries" presenting to a participating level 1 trauma center within 12 hours of their injury, to provide data on the acute post-injury phase. (STUDY COHORT)
- COHORT 2A: Subjects meeting COHORT 2 inclusion criteria, who have UNILATERAL "severe leg injuries". Unilateral injuries include patients who meet the inclusion criteria for a "severe lower extremity injury" for ONE lower extremity, with no more than a simple soft tissue injury (eg, simple laceration) on the contralateral leg.
- COHORT 2B:: Subjects meeting COHORT 2 inclusion criteria, who have BILATERAL lower extremity injuries, with at least one being a "severe leg injury". Bilateral injury patients include patients with at least one lower extremity injury classified as "severe" based on Cohort 2 inclusion criteria, with a contralateral injury greater than a simple soft tissue injury, including femur, foot, and crush injuries. Note that it is not necessary for both lower extremity injuries to meet the inclusion criteria to be enrolled in this cohort.
- COHORT 2C: Subjects meeting COHORT 2 inclusion criteria, clinically diagnosed by the treating provider using that treating provider's standards of diagnosing ACS, and in addition to being diagnosed with ACS, the subject undergoes four-compartment leg fasciotomy. data collection to start BEFORE fasciotomy and continue AFTER fasciotomy.

SUMMARY:
This is a study intended to evaluate a new device that uses light to measure the amount of oxygen in the muscles of injured and non-injured legs and forearms in specific situations. The name of this technology is NIRS (near-infrared spectroscopy). This is a prospective observational cohort study intended to gather data using NIRS among injured and noninjured extremities over time. Additionally, this data will help in establishing diagnostic perfusion value thresholds to be used in a subsequent interventional study confirming the efficacy of NIRS-based ACS monitoring.

DETAILED DESCRIPTION:
Swelling builds up in a severely injured leg (for example, a broken leg). In up to 20% of very bad injuries, the swelling can be so great that it acts to cut off blood supply to the leg, strangulating it from the inside. When this occurs, it is called Acute Compartment Syndrome (ACS). This is a painful and bad situation, which needs to be diagnosed and then surgically treated in an urgent fashion. Currently, the standard way most physicians diagnose ACS is by clinical examination. By asking the patient questions, moving and inspecting the patient's leg and typically inserting a needle in the patient's legs to measure the amount of pressure in each leg. Physicians compile this information and make the final diagnosis. This method of diagnosis can be painful and requires measurements, sometimes invasive, to be made at points in time. ACS is a disease process that develops over time therefore someone may not have ACS at the time of examination, but may develop it several hours later. The treatment for ACS is called a fasciotomy. This treatment involves making a large incision from the knee to the ankle on each side of the lower leg.

The NIRS device has already been cleared by the FDA for detecting blood flow to the brain during anesthesia. NIRS may also be helpful in diagnosing ACS. Two of the primary advantages of this device are that it is noninvasive (not painful) and it collects data continuously, so that if the disease develops, it can be detected early and treated appropriately. In order to prove this, the device must first be tested by taking a series of measurements on people that are uninjured (control groups), those with serious leg injuries (investigational groups), and people in a critically injured state, but without leg injuries (critical controls).

The goal of this study is to collect the information necessary to understand and then create decision-making guidelines that use NIRS monitoring to diagnose and direct treatment for ACS. Information for this study will be collected in the hospital. The study participants will be grouped into 2 categories:

Cohort 1: Patients who are critically injured, but have no lower leg injuries Cohort 2: Patients who have lower leg injuries that fall into certain high-energy categories (see Eligibility Criteria, Section 7.1)

This is an observational study, which means the data collected is not intended to impact the patient's course of care. At all points in time, treatment will be directed by the patient's doctor including decisions regarding operative care, non-operative care and in-patient management. In fact, this study will be blinded, which means that the doctor treating the study patients will not be able to see the NIRS values. This study will enroll approximately 120 subjects over three sites: Athens Regional Medical Center, Atlanta Medical Center, and Grady Memorial Hospital, over a period of approximately 18 months. Participation will last for 48 hours, unless the patient develops signs of compartment syndrome in which case monitoring may be extended up to 72 hours or until completion of an assessment after the patient is treated for ACS.

Participants will undergo the following procedures:

Beyond the standard of care:

1. Patient interview to collect information on medical history, medications, and mechanism of injury
2. Photograph(s) will be taken to document NIRS pad placement over muscle compartments and injury severity (face will not be included).
3. Ultrasound measure of the thickness of the fat layer (BX 2000) to detect the distance from the patient's skin surface to the underlying muscle
4. Light scan measurement of skin color (Dermaspectrometer) to see if the patient's skin color affects NIRS readings
5. Near-infrared Spectroscopy (NIRS) to measure patient's muscle oxygen levels. These devices are completely noninvasive, which means there are no sharp or painful portions of the device or measurement process. The NIRS device uses a small pad, like an EKG pad, that sticks to the patient's skin and gives off a harmless, painless light that can continually measure the patient's muscle oxygen level. These measures are recorded in the monitor and will later be downloaded and used to evaluate the device's ability to detect critical changes in muscle oxygen levels.

Standard of care:

1. Data will be recorded from the patient's medical record based on procedures ordered by the patient's provider, including: lab values, Stryker measurements, vital signs.
2. Among Cohort 2 patients, data associated with some surgical procedures will be collected and recorded in the operating room. This will be data that is gathered as standard of care, such as blood pressure

All of this information will be kept private and secure, and no sensitive information will be collected.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* Admitted to a participating trauma center (Grady, AMC, ARMC) within 12 hours of injury
* At least one uninjured upper extremity
* Patients enrolled in Cohort 2 will have a "severe leg injury" (must be one of the following locations and MOI):

  1. Anatomic Location:
* Tibia/fibula shaft fracture
* Tibial plateau fracture (Schatzker III-VI) 2. High Energy Mechanism of Injury (MOI):
* Fall from >8 foot height
* Motor vehicle collision (>15mph)
* Motor vehicle versus pedestrian accident
* High velocity gunshot wound
* Crush injury
* Sport/recreation
* Patients enrolled in Cohort 1 will meet the criteria listed below:

  1. No bony or vascular lower extremity injury (including femur or foot fractures)
  2. Admitted to the ICU for a traumatic injury (not a medical problem, such as a heart attack)
  3. ICU stay for at least 48 hours(patients with < 2 hours of data will be excluded)

Patients will also be selected for each cohort (See Groups/Cohorts Section).

Exclusion Criteria:

* NIRS monitoring impediment to care
* Known prior leg fractures (not related to current injury)
* Peripheral vascular disease history or concurrent lower extremity vascular injury/surgery
* Admission for medical reasons - atraumatic (ie. myocardial infarction, sepsis…)
* Less 18 years old or greater than 60 years old
* Unable to provide informed consent, or consent cannot be obtained from a legally authorized representative, within 12 hours of injury or prior to first leg surgery, whichever comes first
* Amputation/Mangled Lower Extremity
* Previous fasciotomy history of the injured leg prior to enrollment
* Complete spinal cord injuries
* Bilateral upper extremity injuries
* Participants who are in custody at presentation to the hospital
* Pregnancy
* Open injury on the injured leg that is large enough that at least one NIRS sensor cannot be safely placed over the compartment

  * Spanish-speaking subjects who do not speak English will NOT be excluded. A certified translated copy of the informed consent document will used and a translator will be present for Spanish-speaking patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults who have sustained major blunt and penetrating trauma, who present to Grady Memorial Hospital, Atlanta Medical Center, or Athens Regional Medical Center for treatment meeting the inclusion and exclusion
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
ACS | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Brett Freedman, MD, Principal Investigator — US Army Landstuhl Regional Medical Center
Locations (3):
- United States (3):
  - Athens Regional Medical Center, Athens, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Atlanta Medical Center, Atlanta, Georgia